CLINICAL TRIAL: NCT07245563
Title: Biofilm Formation and Antifungal Resistance in Candida Species: A Comparative Study of Albicans and Non Albicans Strains in Hematology ICU.
Brief Title: Biofilm Formation and Antifungal Resistance in Candida Species
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mennatoallah khaled abdelhady, demonstrator at microbiology department at Assiut university, Assiut University
Other Study IDs: candida species identification
Record Dates: First submitted 2025-10-02; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Candida Infection
MeSH Terms: conditions — Candidiasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — sputum,urine and blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. To determine the susceptibility pattern of our local isolated Candida strains which is essential for optimal management of fungal infection.
2. Detection of biofilm formation by conventional and molecular methods
3. Comparison between C. albicans and non-albicans in the prevalence of biofilm formation and biofilm -forming genes
4. Find the association between antifungal resistance and biofilm formation in candida strains isolated from patients
5. Determination of clinical factors associated with occurrence of infections.

DETAILED DESCRIPTION:
Candida spp are the fourth cause of nosocomial blood stream infections and had a 37% mortality rate within 30-day duration. Early diagnosis of Candida invasive infections reduces the mortality rate from 40% to 15% after therapy .There are several Candida species such as Candida albicans , Candida glabrata but C. albicans remains the most frequent species isolated there is an ongoing shift from C. albicans to non-albicans. Was reported by several countries. C. albicans, C. tropicalis, C. parapsilosis,C. krusei and C. glabrata are responsible for over 90% of cases of candidal infection .Several pathogenic virulence factors are encoded by C. albicans genes and assist the fungus to invade the host tissues leading to infections as the capacity of C. albicans to change from the budding yeast form to filamentous form .Many microbes, including yeasts, form biofilms as one of the major virulence factors. Candida infections often get therapeutic failure, mostly as a result of antifungal resistance that is caused by several mechanisms including biofilm production as biofilm- producing strains show significant increased resistance to antifungal drugs and host immunity.

Candida auris is an emergent pathogen that was first described in Japan. C. auris can be challenging to identify in the laboratory using conventional. Importantly, C. auris isolates are resistant to fluconazole and frequently show multidrug resistance.C. auris has a high capacity for dissemination via contaminated surfaces or horizontal patient-to-patient transfer, which is unusual in other Candida species.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants in the study were those with invasive infection and had one or more of this criteria :

oSuppressed general body immunity.

oSuppressed local body immunity as a result of trauma or invasive procedures.

oResistant to antibiotic therapy.

oNegative samples for bacterial examination and culture.

Critical life threatening infect

Exclusion Criteria:

* Patients who received antifungal therapy within 3 days prior to sample collection.

  * Resistant to antibiotic therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients admitted to hematology intensive care
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-09-20 (Estimated); Study Completion 2026-10-12 (Estimated)

PRIMARY OUTCOMES:
To asses the prevalence of candida species as a cause of infection in patient in hematology intinsive care unit | 1 year
To asses the prevalence of genes responsible for biofilm formation in different candida species | 1 year